CLINICAL TRIAL: NCT05219526
Title: Evaluation of the System Accuracy of 12 Blood Glucose Monitoring Systems According to ISO 15197:2015
Brief Title: System Accuracy of 12 Bloog Glucose Monitoring Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fur Diabetes Karlsburg GmbH (Other)
Collaborators: Aktivmed GmbH (Unknown); Beurer GmbH (Unknown); IME-DC GmbH (Unknown); Medisana GmbH (Unknown)
Responsible Party: Principal Investigator, Matthes Kenning, Director, PhD, Institut fur Diabetes Karlsburg GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IDK_2021_006
Record Dates: First submitted 2021-12-17; First posted 2022-02-02 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject BGMS measurement (Experimental): Blood glucose measurement using BGMS
  Interventions: Diagnostic Test: blood glucose measurement: BGM; Diagnostic Test: blood glucose measurement: reference method

INTERVENTIONS:
Diagnostic Test: blood glucose measurement: BGM — measurement of blood glucose concentration using different BGM
Diagnostic Test: blood glucose measurement: reference method — measurement of blood glucose concentration using reference Method

SUMMARY:
The system accuracy of 12 blood glucose monitoring systems is to be evaluated randomly in accordance with DIN EN ISO 15197:2015 in the course of the year 2022.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with clinical indication for blood glucose measurement
* Signed informed consent form
* Minimum age of 18 years
* Subjects are legally competent and capable to understand character, meaning and consequences of the study.

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with inherent risk of aggravation by the procedure (at the study physician's discretion)
* Current constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* A current constitution that does not allow participating in the study (e.g. hematocrit out of BGM specifications, medication known to influence blood glucose measurements; see Appendix A of ISO 15197)
* Being unable to give informed consent
* < 18 years
* Legally incompetent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement performance: System accuracy | 4-6 hours
  Assessment of the analytical measurement performance of blood glucose monitoring systems based on procedures defined in DIN EN ISO 15197 using results obtained from fingertip blood glucose measurements compared to a reference equipment

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Salzsieder, PhD, Study Director — Institut fur Diabetes Karlsburg GmbH
Locations (1):
- Institut für Diabetes Karlsburg GmbH, Karlsburg, Mecklenburg-Vorpommern, Germany